CLINICAL TRIAL: NCT02861300
Title: Phase I/II Study of CB-839 and Capecitabine in Patients With Advanced Solid Tumors and Fluoropyrimidine Resistant PIK3CA Mutant Colorectal Cancer
Brief Title: CB-839 + Capecitabine in Solid Tumors and Fluoropyrimidine Resistant PIK3CA Mutant Colorectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: David Bajor, MD (Other)
Responsible Party: Sponsor-Investigator, David Bajor, MD, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE1216
Record Dates: First submitted 2016-08-05; First posted 2016-08-10 (Estimated); Results first posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Colorectal Cancer; Colon Cancer; Rectal Cancer; Solid Tumor
Keywords: CB-839; PIK3CA; capecitabine
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Hereditary Sensory and Autonomic Neuropathies | interventions — CB-839; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CB-839 + capecitabine (Experimental): Patients will receive CB-839 orally twice daily for 21 days (continuous administration) and capecitabine orally twice daily for 14/21 days. In the phase I portion of the study, patients will receive escalating doses of CB-839 and capecitabine and will have day 15 blood samples drawn and archived for as needed assessment of CB-839 pharmacokinetics. In the phase II portion of the study, patients will receiving 800mg CB-839 and 1000mg/m^2 capecitabine as were determined to be safe doses during the phase I portion of the study. They will also undergo pre-treatment and post-treatment blood samples and tissue biopsies for evaluation of pharmacodynamic biomarkers.
  Interventions: Drug: CB-839; Drug: Capecitabine

INTERVENTIONS:
Drug: CB-839 — Patients will receive CB-839 orally twice daily during each cycle. Each cycle will be 21 days long. Disease assessment will occur after cycle 3.
Drug: Capecitabine — capecitabine will be given orally twice daily for 14-21 days of cycles. Each cycle will be 21 days long. Disease assessment will occur after cycle 3.
  Other Names: Xeloda

SUMMARY:
This study has two portions. The main goal of the Phase I portion of this research study is to see what doses of CB-839 and capecitabine can safely be given to patients without having too many side effects. Other purposes of this research study will be to determine what side effects are seen with this combination of medicines. The Phase II portion of the study will test how many patients show shrinkage in their tumor with this combination of medicines and what changes occur inside the cancer cells and blood cells after treatment.

DETAILED DESCRIPTION:
Phase I Primary Objective:

To determine the safety, tolerability and recommended phase II dose (RP2D) of combination CB-839 and capecitabine chemotherapy in patients with advanced solid tumors for whom there are no remaining treatment options or for whom single agent capecitabine is an acceptable therapy.

Phase II Primary Objective:

To determine the disease control rate of combination CB-839 and capecitabine chemotherapy in patients with metastatic PIK3CA mutant colorectal cancers who are refractory to fluoropyrimidine based therapy.

Phase I Secondary Objectives:

To determine the dose-limiting toxicities and maximum tolerated dose of combination therapy with CB-839 and capecitabine in patients with advanced solid tumors for whom there are no remaining treatment options or for whom single agent capecitabine is an acceptable therapy.

To determine the disease control rate as assessed by RECIST criteria of combination therapy with CB-839 and capecitabine in patients with advanced solid tumors for whom there are no remaining treatment options or for whom single agent capecitabine is an acceptable therapy.

Phase II Secondary Objectives:

To determine the progression free survival following treatment with CB-839 and capecitabine chemotherapy in patients with metastatic PIK3CA mutant colorectal cancer and are refractory to fluoropyrimidine therapy.

To determine the overall survival following treatment with CB-839 and capecitabine chemotherapy in patients who have metastatic PIK3CA mutant colorectal cancer and are refractory to fluoropyrimidine therapy.

ELIGIBILITY:
Inclusion Criteria:

* Phase I

  * Patients must have an advanced solid tumors for whom there are no remaining treatment options or colorectal patients who have progressed on front-line fluoropyrimidine containing therapy. Patients with colorectal cancer must have progressed on at least one line of fluoropyrimidine containing therapy. Receipt of either oxaliplatin or irinotecan in combination with a fluoropyrimidine is required in the front line setting for all colorectal cancer patients unless either of these agents are otherwise contraindicated in the opinion of the treating physician. Prior regorafenib or TAS-102 therapy is not required.
  * Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
  * Patients must have normal organ and marrow function as defined below:

    * Hemoglobin ≥ 9.0 g/dl
    * Leukocytes ≥ 3,000/mcL
    * Absolute neutrophil count ≥ 1,500/mcL
    * Platelet count ≥ 100,000/mcL
    * Serum creatinine ≤ 1.5 X institutional upper limit of normal
    * Total bilirubin ≤ 1.5mg/dL
    * Aspartate Aminotransferase (AST) serum glutamic oxaloacetic transaminase (SGOT) ≤ 2.5 X institutional upper limit of normal
    * Alanine Aminotransferase (ALT) serum glutamic pyruvic transaminase (SGPT) ≤ 2.5 x institutional upper limit of normal
  * Patients must be able to swallow pills.
  * Patients must have the ability to understand and the willingness to sign a written informed consent document.
  * Female patients of childbearing potential must have a negative serum or urine pregnancy test within 3 days prior to the first dose of study drug and agree to use dual methods of contraception during the study and for a minimum of 3 months following the last dose of study drug. Post-menopausal females (>45 years old and without menses for >1 year) and surgically sterilized females are exempt from these requirements. Male patients must use an effective barrier method of contraception during the study and for a minimum of 3 months following the last dose of study drug if sexually active with a female of childbearing potential.
* Phase II

  * Patients must have histologically or cytologically confirmed, phosphatidylinositol-4,5-bisphosphate 3-kinase catalytic subunit alpha (PIK3CA) mutant metastatic colorectal cancer. PIK3CA status must be confirmed by tumor sequencing in a CLIA certified lab.
  * Patients must have measurable disease according to Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 criteria that is amenable to biopsy and be willing to undergo pre- and post-treatment tumor biopsies. Lesions to be biopsied do not have to be those used for measurement.
  * Patients must have received and progressed on fluoropyrimidine or fluoropyrimidine based therapy. Receipt of either oxaliplatin or irinotecan in combination with a fluoropyrimidine is required in the front line setting unless either of these agents are otherwise contraindicated in the opinion of the treating physician in which case a fluoropyrimidine only may be used. Prior regorafenib or TAS-102 therapy is not required.
  * Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
  * Patients must have normal organ and marrow function as defined below:

    * Hemoglobin ≥ 9.0 g/dl
    * Leukocytes ≥ 3,000/mcL
    * Absolute neutrophil count ≥ 1,500/mcL
    * Platelet count ≥ 100,000/mcL
    * Serum creatinine within normal institutional limits
    * Total bilirubin ≤ 1.5 mg/dL
    * AST (SGOT) ≤ 2.5 X institutional upper limit of normal
    * ALT (SGPT) ≤ 2.5 x institutional upper limit of normal
  * Patients must be able to swallow pills.
  * Patients must have the ability to understand and the willingness to sign a written informed consent document.
  * Female patients of childbearing potential must have a negative serum or urine pregnancy test within 3 days prior to the first dose of study drug and agree to use dual methods of contraception during the study and for a minimum of 3 months following the last dose of study drug. Post-menopausal females (>45 years old and without menses for >1 year) and surgically sterilized females are exempt from these requirements. Male patients must use an effective barrier method of contraception during the study and for a minimum of 3 months following the last dose of study drug if sexually active with a female of childbearing potential.

Exclusion Criteria:

* Both Phase I and Phase II

  * Patients with ongoing toxicities > grade 1 according to National Cancer Institute (NCI) Common Terminology Criteria For Adverse Events (CTCAE) Version 4.0 (excluding alopecia) due to prior anti-cancer therapy.
  * Patients receiving any other investigational agents or whom have received recent treatment for colorectal cancer (radiation within the previous two weeks, chemotherapy or investigational therapy within the previous four weeks).
  * Patients with untreated brain metastases/central nervous system disease will be excluded due to their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
  * Patients with a history of allergic reactions attributed to or intolerance to compounds of similar chemical or biologic composition to either CB-839 or capecitabine. If capecitabine has been received previously, must have tolerated at least an equivalent dose to the dose to be administered at their assigned dose level.
  * Patients who are unable to swallow pills or who have undergone surgery that prohibits the absorption of pills in the stomach.
  * Patients with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris or myocardial infarction within prior 6 months, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
  * Patients who are pregnant or breastfeeding will be excluded from the study.
  * Patients known to be HIV positive who are not receiving anti-retroviral therapy will be excluded due to the marrow suppressive therapy involved in administration of the study treatment.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-09-12 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Bajor, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I Dose -1: * 400 mg CB-839 orally twice daily x 21 days
  * 500 mg/m^2 Capecitabine orally twice daily for 14/21 days
- Phase I Dose 1: * 400 mg CB-839 orally twice daily x 21 days
  * 750 mg/m^2 Capecitabine orally twice daily for 14/21 days
- Phase I Dose 2: * 600 mg CB-839 orally twice daily x 21 days
  * 750 mg/m^2 Capecitabine orally twice daily for 14/21 days
- Phase I Dose 3: * 600 mg CB-839 orally twice daily x 21 days
  * 1000 mg/m^2 Capecitabine orally twice daily for 14/21 days
- Phase I Dose 3A: * 400 mg CB-839 orally twice daily x 21 days
  * 1000 mg/m^2 Capecitabine orally twice daily for 14/21 days
- Phase I Dose 4: * 800 mg CB-839 orally twice daily x 21 days
  * 1000 mg/m^2 Capecitabine orally twice daily for 14/21 days
- Phase II Dose: Recommended Phase I dose of CB-839 and capecitabine
Period: Overall Study
Arm/Group | Phase I Dose -1 | Phase I Dose 1 | Phase I Dose 2 | Phase I Dose 3 | Phase I Dose 3A | Phase I Dose 4 | Phase II Dose
Started | 0 | 3 | 3 | 3 | 0 | 7 | 32
Completed | 0 | 2 | 3 | 3 | 0 | 6 | 3
Not Completed | 0 | 1 | 0 | 0 | 0 | 1 | 29
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 24
Not completed — Delay in treatment | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Disease Progression | 0 | 1 | 0 | 0 | 0 | 0 | 2
Not completed — Patient decision/withdrawal/refusal | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Clinical Complications | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The number of participants analyzed is zero in Phase 1 Dose -1 and Phase 1 Dose 3A because zero participants were enrolled on these arms.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I Dose -1 | Phase I Dose 1 | Phase I Dose 2 | Phase I Dose 3 | Phase I Dose 3A | Phase I Dose 4 | Phase II Dose | Total
Number analyzed (Participants) | 0 | 3 | 3 | 3 | 0 | 7 | 32 | 48
Age, Customized [Count of Participants; unit: Participants] — Rows describe age ranges.
  Participants
    30-39 years of age |  | 0 | 0 | 0 |  | 0 | 3 | 3
    40-49 years of age |  | 1 | 0 | 0 |  | 1 | 4 | 6
    50-59 years of age |  | 1 | 1 | 0 |  | 1 | 13 | 16
    60-69 years of age |  | 0 | 1 | 2 |  | 2 | 10 | 15
    70-79 years of age |  | 1 | 1 | 1 |  | 3 | 3 | 9
    80-89 years of age |  | 0 | 0 | 0 |  | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 2 | 2 | 1 |  | 5 | 18 | 28
  Male |  | 1 | 1 | 2 |  | 2 | 14 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 0 | 0 | 0 |  | 0 | 0 | 0
  Not Hispanic or Latino |  | 3 | 3 | 3 |  | 7 | 31 | 47
  Unknown or Not Reported |  | 0 | 0 | 0 |  | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0 | 0 |  | 0 | 0 | 0
  Asian |  | 0 | 0 | 0 |  | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander |  | 0 | 0 | 0 |  | 0 | 0 | 0
  Black or African American |  | 0 | 0 | 1 |  | 0 | 3 | 4
  White |  | 3 | 3 | 2 |  | 7 | 28 | 43
  More than one race |  | 0 | 0 | 0 |  | 0 | 0 | 0
  Unknown or Not Reported |  | 0 | 0 | 0 |  | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 3 | 3 | 3 |  | 7 | 32 | 48

OUTCOME MEASURES:

1. Primary Outcome: PHASE I: Recommended Dose for Phase II Study
Description: The Phase I study has been designed to define the recommended phase II dose of CB-839 and capecitabine. A traditional 3+3 dose escalation design will be adopted. Nine to twenty-four patients are expected to be enrolled, depending on the number of dose escalations and assuming that a total of 6 patients will be treated at the final recommended phase II dose level. Patients who complete the first 21 day treatment cycle of CB-839 and capecitabine chemotherapy will be included in the analysis.
Time Frame: At least 21 days of treatment
Population: Sixteen participants were enrolled in the Phase I portion of this clinical trial.
Measure: Number; unit: mg/m^2
Groups:
- Phase I: Phase I dose-escalation study of CB-839 and capecitabine in patients with advanced solid tumors and patients for whom single agent capecitabine is an acceptable treatment option.
Arm/Group | Phase I
Number analyzed (Participants) | 16
mg/m^2 | 1,000

2. Primary Outcome: PHASE II: Progression-free Survival (PFS)
Description: The number of participants that achieved PFS will be analyzed. Progression free survival (PFS) on combination CB-839 and capecitabine as determined by clinical assessment and RECIST criteria in patients with metastatic PIK3CA mutant colorectal cancer who are refractory to fluoropyrimidine based therapy. Progression free survival is defined as the time from randomization to documented progression or death without progression.
Time Frame: 6 months
Population: This outcome measure is only relevant to Phase II.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose -1 | Phase I Dose 1 | Phase I Dose 2 | Phase I Dose 3 | Phase I Dose 3A | Phase I Dose 4 | Phase II Dose
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 32
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 7

3. Secondary Outcome: PHASE I: Proportion of Patient Who Respond to Treatment
Description: Disease control rate will be determined using RECIST criteria.
  RECIST response categories: Progressive disease (PD): >=20% increase in sum of longest diameter (LD) of target lesion(s), taking as reference smallest sum LD recorded since treatment started. Complete response (CR): disappearance of all target lesions. Partial response (PR): >=30% decrease in sum of LD of target lesion(s), taking as reference baseline sum LD. Stable disease (SD): neither sufficient shrinkage to qualify as PR nor sufficient increase to qualify as PD.
Time Frame: At least 21 days of treatment
Population: Two participants were not evaluable were are excluded from Phase I Dose 4. This outcome measure only pertains to Phase I therefore Phase II participants are excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose -1 | Phase I Dose 1 | Phase I Dose 2 | Phase I Dose 3 | Phase I Dose 3A | Phase I Dose 4 | Phase II Dose
Number analyzed (Participants) | 0 | 3 | 3 | 3 | 0 | 5 | 0
Participants
  Stable Disease | 0 | 3 | 2 | 3 | 0 | 3 | 0
  Progressive Disease | 0 | 0 | 1 | 0 | 0 | 2 | 0
  Complete Response | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: PHASE I: Dose-limiting Toxicities
Description: Phase I: Dose-limiting toxicities as assessed by CTCAE version 4 of combination CB-839 and capecitabine in patients with advanced solid tumors with no remaining treatment options or patients for whom single agent capecitabine is an acceptable therapy
Time Frame: Up to 18 months after beginning treatment
Population: This outcome measure is only pertaining to Phase I therefore Phase II participants were excluded from the analysis.
Measure: Number; unit: toxicities
Arm/Group | Phase I Dose -1 | Phase I Dose 1 | Phase I Dose 2 | Phase I Dose 3 | Phase I Dose 3A | Phase I Dose 4 | Phase II Dose
Number analyzed (Participants) | 0 | 3 | 3 | 3 | 0 | 7 | 0
toxicities |  | 0 | 0 | 0 |  | 0 |

5. Secondary Outcome: PHASE II: Number of Patients With Response to Treatment
Description: In the phase II component of this study, the primary endpoint is response rate. Disease control rate will be determined using RECIST criteria.
  RECIST response categories: Progressive disease (PD): >=20% increase in sum of longest diameter (LD) of target lesion(s), taking as reference smallest sum LD recorded since treatment started. Complete response (CR): disappearance of all target lesions. Partial response (PR): >=30% decrease in sum of LD of target lesion(s), taking as reference baseline sum LD. Stable disease (SD): neither sufficient shrinkage to qualify as PR nor sufficient increase to qualify as PD.
Time Frame: Up to 18 months after beginning treatment
Population: Only 28 of 32 Phase II participants were evaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose -1 | Phase I Dose 1 | Phase I Dose 2 | Phase I Dose 3 | Phase I Dose 3A | Phase I Dose 4 | Phase II Dose
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 28
Participants
  Stable Disease | 0 | 0 | 0 | 0 | 0 | 0 | 14
  Progressive Disease | 0 | 0 | 0 | 0 | 0 | 0 | 14
  Complete Response | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: PHASE II: Overall Survival
Description: The number of participants to achieve overall survival will be analyzed. Overall survival of patients with metastatic PIK3CA mutant colorectal cancer who are refractory to fluoropyrimidine based therapy following treatment with CB-839 and capecitabine chemotherapy. Overall survival is defined as the time from randomization to death from any cause.
Time Frame: Up to 18 months after beginning treatment
Population: This outcome measure is only relevant to Phase II, therefore no Phase I participants are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose -1 | Phase I Dose 1 | Phase I Dose 2 | Phase I Dose 3 | Phase I Dose 3A | Phase I Dose 4 | Phase II Dose
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 32
Participants |  |  |  |  |  |  | 4

ADVERSE EVENTS:
Time Frame: 18 months after beginning treatment
Description: Arms that enrolled 0 participants have an All-Cause Mortality of zero.
Arm/Group | Phase I Dose -1 | Phase I Dose 1 | Phase I Dose 2 | Phase I Dose 3 | Phase I Dose 3A | Phase I Dose 4 | Phase II Dose
All-Cause Mortality (participants affected / at risk) | 0/0 | 2/3 | 2/3 | 1/3 | 0/0 | 2/7 | 26/32
Serious Adverse Events (participants affected / at risk) | 0/0 | 1/3 | 0/3 | 0/3 | 0/0 | 4/7 | 14/32
Other Adverse Events (participants affected / at risk) | 0/0 | 3/3 | 3/3 | 3/3 | 0/0 | 7/7 | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Dose -1 (N=0) | Phase I Dose 1 (N=3) | Phase I Dose 2 (N=3) | Phase I Dose 3 (N=3) | Phase I Dose 3A (N=0) | Phase I Dose 4 (N=7) | Phase II Dose (N=32)
Hyponatremia (Metabolism and nutrition disorders) | NA | 1 | NA | NA | NA | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | NA | 0 | NA | NA | NA | 1 | 0
Lung Infection (Infections and infestations) | NA | 0 | NA | NA | NA | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | NA | 0 | NA | NA | NA | 1 | 0
Nausea (Gastrointestinal disorders) | NA | 0 | NA | NA | NA | 1 | 4
Vomiting (Gastrointestinal disorders) | NA | 0 | NA | NA | NA | 1 | 4
Abdominal Pain (Gastrointestinal disorders) | NA | 0 | NA | NA | NA | 1 | 2
Skin Infection (Infections and infestations) | NA | 0 | NA | NA | NA | 1 | 0
Anemia (Blood and lymphatic system disorders) | NA | 0 | NA | NA | NA | 0 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | NA | 0 | NA | NA | NA | 0 | 1
Blood bilirubin increased (Investigations) | NA | 0 | NA | NA | NA | 0 | 3
Infections and infestations Other, specify: Cholangitis (Infections and infestations) | NA | 0 | NA | NA | NA | 0 | 1
Colonic obstruction (Gastrointestinal disorders) | NA | 0 | NA | NA | NA | 0 | 1
Creatinine increased (Investigations) | NA | 0 | NA | NA | NA | 0 | 2
Death NOS (General disorders) | NA | 0 | NA | NA | NA | 0 | 1
Diarrhea (Gastrointestinal disorders) | NA | 0 | NA | NA | NA | 0 | 3
Infections and infestations Other, specify: Diverticulitis (Infections and infestations) | NA | 0 | NA | NA | NA | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | NA | 0 | NA | NA | NA | 0 | 2
Fatigue (General disorders) | NA | 0 | NA | NA | NA | 0 | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | NA | 0 | NA | NA | NA | 0 | 3
Gastroesophageal reflux disease (Gastrointestinal disorders) | NA | 0 | NA | NA | NA | 0 | 1
Hematuria (Renal and urinary disorders) | NA | 0 | NA | NA | NA | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | NA | 0 | NA | NA | NA | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | NA | 0 | NA | NA | NA | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | NA | 0 | NA | NA | NA | 0 | 1
Depression (Psychiatric disorders) | NA | 0 | NA | NA | NA | 0 | 1
Sepsis (Infections and infestations) | NA | 0 | NA | NA | NA | 0 | 2
General disorders and administration site conditions Other, specify: Lactic Acidosis (General disorders) | NA | 0 | NA | NA | NA | 0 | 1
Hepatobiliary disorders - Other, specify: Malignant Biliary Obstruction (Hepatobiliary disorders) | NA | 0 | NA | NA | NA | 0 | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | NA | 0 | NA | NA | NA | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | NA | 0 | NA | NA | NA | 0 | 1
Skin infection (Infections and infestations) | NA | 0 | NA | NA | NA | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | NA | 0 | NA | NA | NA | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Dose -1 (N=0) | Phase I Dose 1 (N=3) | Phase I Dose 2 (N=3) | Phase I Dose 3 (N=3) | Phase I Dose 3A (N=0) | Phase I Dose 4 (N=7) | Phase II Dose (N=32)
Abdominal distention (Gastrointestinal disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Abdominal pain (Gastrointestinal disorders) | NA | 0 | 0 | 0 | NA | 0 | 11
Acute kidney injury (Renal and urinary disorders) | NA | 1 | 0 | 0 | NA | 0 | 1
Akathisia (Nervous system disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Alanine aminotransferase increased (Investigations) | NA | 0 | 2 | 2 | NA | 1 | 12
Alkaline phosphatase increased (Investigations) | NA | 1 | 0 | 2 | NA | 3 | 11
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | NA | 1 | 0 | 0 | NA | 1 | 1
Anemia (Blood and lymphatic system disorders) | NA | 1 | 1 | 2 | NA | 5 | 15
Anorexia (Metabolism and nutrition disorders) | NA | 0 | 2 | 1 | NA | 2 | 12
Anxiety (Psychiatric disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | NA | 0 | 0 | 0 | NA | 0 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Aspartate aminotransferase increased (Investigations) | NA | 0 | 2 | 2 | NA | 2 | 16
Aspiration (Respiratory, thoracic and mediastinal disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Atrial Fibrillation (Cardiac disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | NA | 0 | 0 | 0 | NA | 0 | 5
Bladder Spasm (Renal and urinary disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Bloating (Gastrointestinal disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Blood and lymphatic system disorders- Other, specify: Low serum Vitamin D (Blood and lymphatic system disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Blood bilirubin increased (Investigations) | NA | 0 | 1 | 2 | NA | 4 | 11
Blurred Vision (Eye disorders) | NA | 0 | 0 | 0 | NA | 1 | 4
Bullous dermatitis (Skin and subcutaneous tissue disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Chills (General disorders) | NA | 1 | 0 | 0 | NA | 0 | 4
Cholecystitis (Hepatobiliary disorders) | NA | 0 | 0 | 0 | NA | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Concentration impairment (Nervous system disorders) | NA | 0 | 0 | 0 | NA | 0 | 3
Constipation (Gastrointestinal disorders) | NA | 0 | 1 | 1 | NA | 3 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | NA | 0 | 0 | 0 | NA | 2 | 1
Creatinine increased (Investigations) | NA | 2 | 0 | 0 | NA | 3 | 6
Cystitis noninfective (Renal and urinary disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Dehydration (Metabolism and nutrition disorders) | NA | 0 | 0 | 0 | NA | 1 | 5
Depression (Psychiatric disorders) | NA | 0 | 0 | 1 | NA | 0 | 2
Diarrhea (Gastrointestinal disorders) | NA | 1 | 0 | 0 | NA | 3 | 14
Dizziness (Nervous system disorders) | NA | 0 | 1 | 0 | NA | 1 | 3
Dry eye (Eye disorders) | NA | 0 | 0 | 1 | NA | 0 | 2
Dry mouth (Gastrointestinal disorders) | NA | 0 | 0 | 0 | NA | 0 | 4
Dry skin (Skin and subcutaneous tissue disorders) | NA | 1 | 0 | 0 | NA | 0 | 3
Dysgeusia (Nervous system disorders) | NA | 0 | 0 | 0 | NA | 1 | 7
Dyspepsia (Gastrointestinal disorders) | NA | 0 | 0 | 0 | NA | 1 | 0
Dysphagia (Gastrointestinal disorders) | NA | 0 | 0 | 0 | NA | 0 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | NA | 1 | 0 | 1 | NA | 2 | 2
Ear and labyrinth disorders Other, specify: Ear congestion (Ear and labyrinth disorders) | NA | 1 | 0 | 0 | NA | 0 | 0
Edema Limbs (General disorders) | NA | 0 | 0 | 0 | NA | 4 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Esophageal Pain (Gastrointestinal disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Eye disorder - Other, specify: brighter light around perimeter of vision (Eye disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Eye disorder - Other, specify: Eye heaviness (Eye disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Eye disorders - Other, specify: Bilateral eye crusting (Eye disorders) | NA | 1 | 0 | 0 | NA | 0 | 0
Eye disorders - Other, specify: NOS (Eye disorders) | NA | 0 | 0 | 0 | NA | 0 | 2
Eye disorders - Other, specify: Right eye pruritis (Eye disorders) | NA | 1 | 0 | 0 | NA | 0 | 0
Eye disorders - Other, specify: Visual auras (Eye disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Eye pain (Eye disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Fall (Injury, poisoning and procedural complications) | NA | 1 | 0 | 1 | NA | 0 | 1
Fatigue (General disorders) | NA | 1 | 2 | 1 | NA | 3 | 17
Fever (General disorders) | NA | 0 | 0 | 0 | NA | 0 | 4
Flank pain (Musculoskeletal and connective tissue disorders) | NA | 0 | 0 | 0 | NA | 0 | 3
Flashing lights (Eye disorders) | NA | 1 | 0 | 0 | NA | 0 | 0
Flatulence (Gastrointestinal disorders) | NA | 0 | 0 | 0 | NA | 1 | 1
Fracture (Injury, poisoning and procedural complications) | NA | 0 | 0 | 1 | NA | 0 | 0
Gait Disturbance (General disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Gastrointestinal disorders - Other, specify: Tenesmus (Gastrointestinal disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Gastrointestinal disorders Other, specify- Mouth Sore (Gastrointestinal disorders) | NA | 2 | 0 | 0 | NA | 0 | 0
Gastrointestinal disorders- Other, specify: Hard stool (Gastrointestinal disorders) | NA | 0 | 0 | 0 | NA | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | NA | 0 | 0 | 0 | NA | 0 | 3
General disorders and administration site conditions Other, Specify- Laceration (General disorders) | NA | 1 | 0 | 0 | NA | 0 | 0
General disorders and administration site conditions Other, Specify- Lower left quadrant pain (General disorders) | NA | 0 | 1 | 0 | NA | 0 | 0
General disorders and administration site conditions- Other, specify: biopsy site pain (General disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
General disorders and administration site conditions- Other, specify: Body Aches (General disorders) | NA | 1 | 0 | 0 | NA | 0 | 0
General disorders and administration site conditions- Other, specify: Generalized Weakness (General disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
General disorders and administration site conditions- Other,specify:ankle swelling (General disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
General disorders and administration site conditions: other, specify: Cold Symptoms (General disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | NA | 0 | 0 | 0 | NA | 3 | 5
Headache (Nervous system disorders) | NA | 0 | 0 | 0 | NA | 0 | 5
Hematuria (Renal and urinary disorders) | NA | 1 | 1 | 0 | NA | 0 | 1
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | NA | 0 | 1 | 0 | NA | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | NA | 0 | 0 | 0 | NA | 0 | 2
Hot flashes (Vascular disorders) | NA | 0 | 0 | 0 | NA | 1 | 2
Hypercalcemia (Metabolism and nutrition disorders) | NA | 0 | 1 | 0 | NA | 1 | 2
Hyperglycemia (Metabolism and nutrition disorders) | NA | 0 | 1 | 0 | NA | 0 | 11
Hyperkalemia (Metabolism and nutrition disorders) | NA | 0 | 1 | 1 | NA | 0 | 1
hypermagnesemia (Metabolism and nutrition disorders) | NA | 2 | 0 | 0 | NA | 0 | 2
Hypertension (Metabolism and nutrition disorders) | NA | 0 | 1 | 0 | NA | 3 | 7
Hypoalbuminemia (Metabolism and nutrition disorders) | NA | 0 | 1 | 0 | NA | 5 | 8
Hypocalcemia (Metabolism and nutrition disorders) | NA | 0 | 0 | 0 | NA | 1 | 5
Hypochloremia (Metabolism and nutrition disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | NA | 2 | 0 | 0 | NA | 1 | 2
Hypokalemia (Metabolism and nutrition disorders) | NA | 0 | 0 | 0 | NA | 4 | 10
Hypomagnesemia (Metabolism and nutrition disorders) | NA | 1 | 1 | 2 | NA | 2 | 8
Hyponatremia (Metabolism and nutrition disorders) | NA | 3 | 3 | 2 | NA | 3 | 14
Hypophosphatemia (Investigations) | NA | 0 | 0 | 1 | NA | 4 | 11
Hypotension (Metabolism and nutrition disorders) | NA | 0 | 0 | 0 | NA | 0 | 2
Hypoxia (Metabolism and nutrition disorders) | NA | 0 | 0 | 0 | NA | 1 | 0
Infections and infestations Other, specify: Cold sore (Infections and infestations) | NA | 1 | 0 | 0 | NA | 0 | 0
Infections and infestations Other, specify: Oral thrush (Infections and infestations) | NA | 0 | 0 | 0 | NA | 1 | 0
Injury, poisoning and procedural complications - Other, specify: NOS (Injury, poisoning and procedural complications) | NA | 0 | 0 | 0 | NA | 0 | 1
INR increased (Investigations) | NA | 0 | 0 | 0 | NA | 2 | 3
Insomnia (Psychiatric disorders) | NA | 0 | 1 | 0 | NA | 1 | 2
Intestinal stoma site bleeding (Injury, poisoning and procedural complications) | NA | 0 | 0 | 0 | NA | 0 | 1
Investigations - Other, specify: Alkaline phosphatase decreased (Investigations) | NA | 0 | 0 | 0 | NA | 0 | 1
Investigations - Other, specify: Low cholesterol (Investigations) | NA | 0 | 0 | 0 | NA | 0 | 1
Investigations - Other, specify: Low Creatinine (Investigations) | NA | 0 | 0 | 0 | NA | 0 | 1
Investigations - Other, specify: Monocyte Count Elevated (Investigations) | NA | 0 | 0 | 0 | NA | 0 | 1
Investigations- Other, specify: Decreased Anion Gap (Investigations) | NA | 0 | 0 | 0 | NA | 0 | 1
Investigations- Other, Specify: Elevated blood urea nitrogen (Investigations) | NA | 0 | 0 | 0 | NA | 0 | 1
Investigations- Other, Specify: Hyperchloremia (Investigations) | NA | 0 | 0 | 0 | NA | 0 | 1
Lethargy (Nervous system disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | NA | 0 | 0 | 0 | NA | 1 | 2
Lipase increased (Investigations) | NA | 0 | 0 | 0 | NA | 0 | 1
Lymph Node Pain (Blood and lymphatic system disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Lymphedema (Vascular disorders) | NA | 0 | 0 | 0 | NA | 1 | 1
Lymphocyte count decreased (Investigations) | NA | 3 | 1 | 1 | NA | 6 | 14
Malaise (General disorders) | NA | 0 | 0 | 0 | NA | 1 | 1
Menorrhagia (Reproductive system and breast disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Metabolism and nutrition disorders: other, specify- decreased appetite (Metabolism and nutrition disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Mucositis oral (Gastrointestinal disorders) | NA | 0 | 0 | 0 | NA | 1 | 8
Musculoskeletal and connective tissue disorder - Other, specify: Pseudogout (Musculoskeletal and connective tissue disorders) | NA | 0 | 0 | 0 | NA | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | NA | 0 | 0 | 0 | NA | 1 | 0
Nail discoloration (Skin and subcutaneous tissue disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Nail infection (Infections and infestations) | NA | 0 | 0 | 1 | NA | 0 | 0
Nail loss (Skin and subcutaneous tissue disorders) | NA | 0 | 0 | 1 | NA | 1 | 1
Nail ridging (Skin and subcutaneous tissue disorders) | NA | 0 | 0 | 1 | NA | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | NA | 0 | 1 | 0 | NA | 0 | 2
Nausea (Gastrointestinal disorders) | NA | 1 | 1 | 1 | NA | 4 | 18
Neck pain (Musculoskeletal and connective tissue disorders) | NA | 0 | 0 | 0 | NA | 0 | 2
Nervous system disorders - Other, specify: NOS (Nervous system disorders) | NA | 0 | 0 | 0 | NA | 1 | 0
Nervous system disorders- Other, specify: Increased area of neuropathy (Nervous system disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Nervous system disorders: Other, specify- Neuropathic Extremity (Nervous system disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Neuralgia (Nervous system disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Neutrophil count decreased (Investigations) | NA | 0 | 0 | 0 | NA | 1 | 1
Non-cardiac chest pain (General disorders) | NA | 0 | 0 | 0 | NA | 1 | 3
Oral dysesthesia (Gastrointestinal disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Pain (General disorders) | NA | 1 | 3 | 1 | NA | 4 | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | NA | 1 | 1 | 1 | NA | 1 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | NA | 2 | 1 | 1 | NA | 5 | 13
Palpitations (Cardiac disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Papulopustular rash (Infections and infestations) | NA | 0 | 0 | 0 | NA | 0 | 1
Paresthesia (Nervous system disorders) | NA | 0 | 0 | 0 | NA | 0 | 3
Pelvic Pain (Reproductive system and breast disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | NA | 0 | 0 | 0 | NA | 1 | 4
Photophobia (Eye disorders) | NA | 2 | 2 | 3 | NA | 4 | 4
Photosensitivity (Skin and subcutaneous tissue disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Platelet count decreased (Investigations) | NA | 1 | 0 | 2 | NA | 4 | 5
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Prolapse of intestinal stoma (Injury, poisoning and procedural complications) | NA | 0 | 0 | 0 | NA | 0 | 1
Proteinuria (Renal and urinary disorders) | NA | 1 | 0 | 0 | NA | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | NA | 0 | 0 | 0 | NA | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Rectal hemorrhage (Gastrointestinal disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Rectal pain (Gastrointestinal disorders) | NA | 1 | 0 | 0 | NA | 0 | 1
Renal and urinary disorders - Other, specify: NOS (Renal and urinary disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Renal and urinary disorders- Other, specify: Urinary hesitancy (Renal and urinary disorders) | NA | 0 | 0 | 0 | NA | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify: Sinus Drainage (Respiratory, thoracic and mediastinal disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Sinus bradycardia (Cardiac disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Sinus tachycardia (Cardiac disorders) | NA | 0 | 0 | 0 | NA | 1 | 0
Skin and subcutaneous tissue disorders - Other, specify: cracked skin in corner of mouth (Skin and subcutaneous tissue disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Skin and subcutaneous tissue disorders - Other, specify: Finger cut (Skin and subcutaneous tissue disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Skin and subcutaneous tissue disorders - Other, specify: NOS (Skin and subcutaneous tissue disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Skin and subcutaneous tissue disorders - Other, specify: Rash to Chest, Neck (occasional pruritus) (Skin and subcutaneous tissue disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Skin and subcutaneous tissue disorders - Other, specify: Rash to Chest and Neck-No Pruritis/No Pain (Skin and subcutaneous tissue disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Skin and subcutaneous tissue disorders - Other, specify: Skin Discoloration (Skin and subcutaneous tissue disorders) | NA | 0 | 0 | 1 | NA | 0 | 0
Skin and subcutaneous tissue disorders - Other, specify: two small red spots on her right cheek (Skin and subcutaneous tissue disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Skin and subcutaneous tissue disorders- Other, Specify: Brittle Nails (Skin and subcutaneous tissue disorders) | NA | 0 | 0 | 0 | NA | 1 | 0
Skin and subcutaneous tissue disorders- Other, specify: Sores on body (Skin and subcutaneous tissue disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Skin and subcutaneous tissue disorders- Other, specify: Swelling around bilateral big toe nails (Skin and subcutaneous tissue disorders) | NA | 1 | 0 | 0 | NA | 0 | 0
Skin and subcutaneous tissue disorders: Other, specify- Inflammation of Actinic Keratosis (Skin and subcutaneous tissue disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Skin and subcutaneous tissue disorders: Other, specify: Intertrigo (Skin and subcutaneous tissue disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Skin induration (Skin and subcutaneous tissue disorders) | NA | 0 | 0 | 0 | NA | 1 | 0
Skin Infection (Infections and infestations) | NA | 0 | 1 | 0 | NA | 0 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Somnolence (Nervous system disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | NA | 1 | 0 | 0 | NA | 0 | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | 0 | 0 | 0 | NA | 0 | 1
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Urinary fistula (Renal and urinary disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Urinary frequency (Renal and urinary disorders) | NA | 1 | 0 | 0 | NA | 0 | 2
Urinary incontinence (Renal and urinary disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Urinary retention (Renal and urinary disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Urinary Tract Infection (Renal and urinary disorders) | NA | 1 | 0 | 0 | NA | 1 | 3
Urinary tract pain (Renal and urinary disorders) | NA | 0 | 0 | 1 | NA | 0 | 1
Urine Discoloration (Renal and urinary disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Vaginal Dryness (Reproductive system and breast disorders) | NA | 1 | 0 | 0 | NA | 0 | 0
Vaginal hemorrhage (Reproductive system and breast disorders) | NA | 1 | 0 | 0 | NA | 0 | 0
Vaginal Pain (Reproductive system and breast disorders) | NA | 1 | 0 | 0 | NA | 0 | 1
Vascular disorders- Other, specify: Broken capillaries at skin surface (Vascular disorders) | NA | 0 | 0 | 0 | NA | 0 | 1
Vomiting (Gastrointestinal disorders) | NA | 1 | 1 | 0 | NA | 6 | 9
Watering eyes (Eye disorders) | NA | 0 | 0 | 1 | NA | 0 | 2
Weight gain (Investigations) | NA | 0 | 0 | 0 | NA | 1 | 0
Weight Loss (Investigations) | NA | 0 | 1 | 1 | NA | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | NA | 0 | 0 | 0 | NA | 0 | 3
White blood cell decreased (Investigations) | NA | 3 | 1 | 1 | NA | 3 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-16): https://cdn.clinicaltrials.gov/large-docs/00/NCT02861300/Prot_SAP_000.pdf
  • Informed Consent Form (2023-10-25): https://cdn.clinicaltrials.gov/large-docs/00/NCT02861300/ICF_001.pdf